CLINICAL TRIAL: NCT02320695
Title: Evaluation of Perception of Sting Sensation Following Application of Antibiotic Ointment and Cream Formulations After Tape Stripping Injury
Brief Title: Trial to Test if Antibiotic Ointments & Cream Will Sting After Application on a Minor Wound After Tape Stripping Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CO-140617115421-THCT
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Sting
MeSH Terms: conditions — Bites and Stings | interventions — Sodium Chloride; 2-Propanol; bacitracin zinc, neomycin sulfate, polymyxin B, drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Saline (Placebo Comparator): 0.9% Sodium Chloride Saline Solution (0.3 cc)
  Interventions: Drug: Saline
- Isopropyl Alcohol (Placebo Comparator): 70% Isopropyl Alcohol (0.3 cc)
  Interventions: Drug: Isopropyl Alcohol
- Pain Relieving Cream (Experimental): Neosporin® Plus Pain Relieving Cream formula with pH balance technology (0.3 cc)
  Interventions: Drug: Pain Relieving Cream
- Antibiotic/Pain Relieving Ointment (Experimental): Neosporin® Complete First Aid Antibiotic/Pain Relieving Ointment (0.3 cc)
  Interventions: Drug: Antibiotic/Pain Relieving Ointment
- Original Ointment (Experimental): Neosporin® Original Ointment (0.3 cc)
  Interventions: Drug: Original Ointment
- Pain Relief Ointment (Experimental): Neosporin® Plus Pain relief Ointment (0.3 cc)
  Interventions: Drug: Pain Relief Ointment

INTERVENTIONS:
Drug: Saline
  Other Names: Sterile 0.9% Sodium Chloride Saline Solution
  Arms: Saline
Drug: Isopropyl Alcohol
  Other Names: 70 % Isopropyl Alcohol
  Arms: Isopropyl Alcohol
Drug: Pain Relieving Cream
  Other Names: Neosporin® Plus Pain Relieving Cream formula with pH balance technology
  Arms: Pain Relieving Cream
Drug: Antibiotic/Pain Relieving Ointment
  Other Names: Neosporin® Complete First Aid Antibiotic/Pain Relieving Ointment
  Arms: Antibiotic/Pain Relieving Ointment
Drug: Original Ointment
  Other Names: Neosporin® Original Ointment
  Arms: Original Ointment
Drug: Pain Relief Ointment
  Other Names: Neosporin® Plus Pain relief Ointment
  Arms: Pain Relief Ointment

SUMMARY:
The purpose of this study is to have subjects report whether or not several antibiotic products sting when they are applied to minor wounds created on the inner arms.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the sting potential of single applications of over-the-counter (OTC) topical antibiotic ointments and cream compared to saline (negative control) and isopropyl alcohol (positive control) when applied to a tape-stripped wound site.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-75 years of age, of any race or ethnicity, in generally good health as determined by a medically-qualified individual
2. Provide a signed and dated informed consent form prior to start of any study-related procedures
3. Able to comprehend and follow the requirements of the study;
4. Females of childbearing potential must have a negative urine pregnancy test at the Screening/Baseline visit;
5. Male or non-pregnant, non-lactating females agree to the contraceptive requirements (including female partner's use of a highly effective form of birth control. Females must have used the same birth control for 1 month before Screening and continue to use it through 1 month after administration of study drug)
6. Willing and able to comply with the tape stripping and all study procedures and attend the scheduled visits for the duration of the study

Exclusion Criteria:

1. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates)
2. Females who are pregnant (positive urine pregnancy test at screening/baseline) or breastfeeding
3. Males with a pregnant partner or a partner who is currently trying to become pregnant
4. Using steroidal medication (topical or systemic) currently and within 30 days before Visit 1
5. Ingestion of systemic anti-histamines or analgesics within the 3 days before Visit 1
6. Known sensitivity or allergies to the investigational products, to first aid preparations or local anesthetics (e.g. gauze products, pramoxine), or to adhesive bandages
7. Known allergies to unscented soap
8. Tendency of forming keloids after wounding
9. Tattoos located on the surface of one or both inner (volar) region of forearms
10. Heavily pigmented subjects who could heal with abnormal darkening at the test sites on the inner forearms
11. Presence of excessive hair on the inner forearms which could interfere with the test procedures
12. Presents with skin disorders on the inner arms (cuts, scratches, scars, etc), which in the opinion of the Investigator or qualified designee, will interfere with the study assessment or will create undue risk for the subject
13. Pre-existing or dormant dermatologic skin conditions (e.g., eczema, seborrheic dermatitis, atopic dermatitis, psoriasis, vitiligo, etc.) that could interfere with the outcome of the study as determined by the Investigator or qualified designee
14. Other medical condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nunez, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide

RESULTS

PARTICIPANT FLOW:
Groups:
- OVERALL: Subjects were assigned to each of the following interventions: Saline, Isopropyl Alcohol, Neosporin Plus Pain Relieving Cream, Neosporin Complete First Aid Antibiotic/Pain Relieving Ointment, Neosporin Original Ointment, Neosporin Plus Pain Relief Ointment. The sequence in which participants received the intervention was randomized.
Period: Overall Study
Arm/Group | OVERALL
Started | 60
Saline | 60
Alcohol | 60
Pain Relieving Cream | 59
Antibiotic/Pain Relieving Ointment | 60
Original Ointment | 60
Pain Relief Ointment | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- OVERALL: This includes all 60 randomized subjects. Subjects were assigned to each of the following interventions: Saline, Isopropyl Alcohol, Neosporin Plus Pain Relieving Cream, Neosporin Complete First Aid Antibiotic/Pain Relieving Ointment, Neosporin Original Ointment, Neosporin Plus Pain Relief Ointment. The sequence in which participants received the intervention was randomized.
Arm/Group | OVERALL
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Post-Tape Stripping in Subject Assessment of Stinging Sensation Immediately After Investigational Product Application
Description: The stinging sensation was assessed by the subject using the following scale: 0 = no stinging sensation, 1 = mild stinging sensation, 2 = moderate stinging sensation, and 3 = severe stinging sensation at post-tape stripping and immediately after product application. Change from post-tape striping was calculated as the subject assessment of stinging sensation immediately after investigational product application minus the subject assessment of stinging sensation at post-tape stripping.
Time Frame: Post-tape stripping to immediately after investigational product application
Population: Analysis was based on all randomized subjects who initiated the tape-stripping procedures and perceived sting sensation immediately after the application of alcohol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Isopropyl Alcohol | Pain Relieving Cream | Antibiotic/Pain Relieving Ointment | Original Ointment | Pain Relief Ointment
Number analyzed (Participants) | 34 | 34 | 33 | 34 | 34 | 34
units on a scale | -0.29 (0.84) | 0.82 (0.94) | -0.55 (0.67) | -0.65 (0.73) | -0.47 (0.61) | -0.71 (0.58)
Statistical Analysis 1: Comparison: Saline vs Pain Relieving Cream; Test type: Non-Inferiority or Equivalence — For the purpose of showing "equivalent stinging" of investigational product to saline, the hypothesis was set up as: Ho: μ1 - μ2 ≥ D vs HA: μ1 - μ2 < D where D was the non-inferiority margin. "Equivalent stinging" of investigational product to saline was claimed if the upper limit of the two-sided 95% confidence interval of (investigational product - saline) was less than 0.5; p = 0.187, ANCOVA; Terms included treatment as factor, post tape-stripping score as covariate and subject as random effect to incorporate within-subject correlations; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.33 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Saline vs Antibiotic/Pain Relieving Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.101, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.42 to 0.04], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Saline vs Original Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.49 to -0.10], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Saline vs Pain Relief Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.53 to -0.12], Standard Error of Mean 0.12

2. Primary Outcome: Mean Change From Post-Tape Stripping in Subject Assessment of Stinging Sensation One Minute After Investigational Product Application
Description: The stinging sensation was assessed by the subject using the following scale: 0 = no stinging sensation, 1 = mild stinging sensation, 2 = moderate stinging sensation, and 3 = severe stinging sensation at post-tape stripping and one minute after investigational product application. Change from post-tape striping was calculated as the subject assessment of stinging sensation at one minute after investigational product application minus the subject assessment of stinging sensation at post-tape stripping.
Time Frame: Post-tape stripping to one minute after investigational product application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Isopropyl Alcohol | Pain Relieving Cream | Antibiotic/Pain Relieving Ointment | Original Ointment | Pain Relief Ointment
Number analyzed (Participants) | 34 | 34 | 33 | 34 | 34 | 34
units on a scale | -0.24 (0.92) | -0.35 (0.73) | -0.67 (0.65) | -0.47 (0.86) | -0.50 (0.56) | -0.68 (0.64)
Statistical Analysis 1: Comparison: Saline vs Pain Relieving Cream; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.023, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.29, 95% CI 2-sided [-0.54 to -0.05], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Saline vs Antibiotic/Pain Relieving Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.522, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.32 to 0.20], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Saline vs Original Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.67 to -0.16], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Saline vs Pain Relief Ointment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.013, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.63 to -0.07], Standard Error of Mean 0.12

3. Secondary Outcome: Mean Clinician Rating of Overall Wound Condition on Day 1
Description: The clinician evaluated the wound using the following scale: 0 = minimal severity, 10 = maximal severity.
Time Frame: Day 1
Population: The Intent-to-Treat (ITT) analysis population included all randomized subjects who had initiated the tape-stripping procedures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Isopropyl Alcohol | Pain Relieving Cream | Antibiotic/Pain Relieving Ointment | Original Ointment | Pain Relief Ointment
Number analyzed (Participants) | 60 | 60 | 59 | 60 | 60 | 60
units on a scale | 2.42 (1.18) | 2.10 (1.02) | 2.22 (1.00) | 2.50 (1.13) | 2.32 (1.23) | 2.15 (0.97)

4. Secondary Outcome: Mean Clinician Rating of Overall Wound Condition on Day 8
Description: The clinician evaluated the wound using the following scale: 0 = minimal severity, 10 = maximal severity.
Time Frame: Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Isopropyl Alcohol | Pain Relieving Cream | Antibiotic/Pain Relieving Ointment | Original Ointment | Pain Relief Ointment
Number analyzed (Participants) | 60 | 60 | 59 | 60 | 60 | 60
units on a scale | 1.43 (0.85) | 1.35 (0.68) | 1.37 (0.83) | 1.35 (0.73) | 1.47 (0.89) | 1.38 (0.76)

ADVERSE EVENTS:
Time Frame: Approximately seven days, +30 days for serious adverse events.
Description: Adverse events were systematically collected on Study Day 1 (Visit 1) and approximately seven days later at the end of study visit (Visit 2). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Groups:
- OVERALL: This includes all 60 randomized subjects.
Arm/Group | OVERALL
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.